CLINICAL TRIAL: NCT07264803
Title: A Single-arm Clinical Trial Using Patient-derived Tumor Tissue Fragment Models for Drug Sensitivity Testing to Guide Treatment in Refractory Cancers
Brief Title: A Single-arm Clinical Trial Using Patient-derived Tumor Tissue Fragment Models for Drug Sensitivity Testing to Guide Treatment in Previously Treated Cancers
Acronym: PDTF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Lian Liu, MD, PHD, Professor and Director, Department of Oncology, Qilu Hospital of Shandong University, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDTF
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor Malignancies; Solid Tumor Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PDTF-Guided Personalized Treatment Arm (Experimental): Patients with refractory solid tumors will undergo drug sensitivity testing using patient-derived tumor tissue fragment (PDTF) models. Fresh tumor tissues obtained from biopsy or surgery will be processed to establish PDTF models that preserve the original tumor microenvironment. Each PDTF will be exposed ex vivo to a panel of anti-cancer agents, including chemotherapy drugs, targeted agents, or immunotherapy drugs.
  Based on the PDTF drug response profiles, an individualized treatment regimen will be formulated after obtaining sensitivity results. Patients will then receive the PDTF-guided regimen until disease progression, unacceptable toxicity, or withdrawal. The effectiveness of the PDTF-guided therapy will be evaluated by tumor response, disease control, and survival outcomes.
  Interventions: Other: PDTF-Guided Personalized Treatment

INTERVENTIONS:
Other: PDTF-Guided Personalized Treatment — Patients with refractory solid tumors in this arm will undergo drug sensitivity testing using patient-derived tumor tissue fragment (PDTF) models. Fresh tumor tissues obtained from biopsy or surgery will be processed to establish PDTF models that preserve the original tumor architecture and microenvironment. Each PDTF will be exposed ex vivo to a panel of anti-cancer agents, including chemotherapy, targeted therapies, and/or immunotherapy drugs.
  Based on the PDTF drug response profiles, an individualized treatment regimen will be formulated after obtaining the sensitivity results. Patients will then receive the PDTF-guided regimen until disease progression, unacceptable toxicity, death, or withdrawal of consent. Clinical outcomes and concordance between PDTF sensitivity and in-vivo treatment response will be assessed.
Other: PDTF-Guided Personalized Treatment — Patients with refractory solid tumors in this arm will undergo drug sensitivity testing using patient-derived tumor tissue fragment (PDTF) models. Fresh tumor tissues obtained from biopsy or surgery will be processed to establish PDTF models that preserve the original tumor architecture and microenvironment. Each PDTF will be exposed ex vivo to a panel of guideline-recommended, FDA- or NMPA-approved anti-cancer agents, including chemotherapy, targeted therapies, and/or immunotherapy drugs.
  Based on the PDTF drug response profiles, an individualized treatment regimen will be formulated within 24 hours after obtaining the sensitivity results. Patients will then receive the PDTF-guided regimen until disease progression, unacceptable toxicity, death, or withdrawal of consent. Clinical outcomes and concordance between PDTF sensitivity and in-vivo treatment response will be assessed.

SUMMARY:
This is a prospective, single-arm, open-label, exploratory clinical trial conducted at Qilu Hospital of Shandong University. Approximately 35 patients with advanced or metastatic refractory cancers will be enrolled. Fresh tumor or metastatic biopsy samples will be collected to establish patient-derived tumor tissue fragment models (PDTFs). Each PDTF will be validated for histologic, molecular, and genetic homology with the original tumor, followed by high-throughput ex vivo drug sensitivity testing using chemotherapy, targeted agents, or immunotherapy drugs and recommended by clinical guidelines.

This study aims to demonstrate that the PDTF platform can serve as a rapid, reliable, and clinically relevant tool for precision therapy development and clinical decision-making in refractory cancers, potentially bridging translational models and individualized clinical care.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following criteria simultaneously to be eligible for enrollment. All criteria must be confirmed through clinical evaluation, laboratory tests, and imaging during the screening period, and approved in writing by the principal investigator.

1. Age between 18 and 75 years (inclusive), regardless of gender.
2. Confirmed diagnosis of refractory malignant tumors via pathological biopsy, including locally advanced unresectable or metastatic gastric cancer or gastroesophageal junction adenocarcinoma; confirmed as stage IV (advanced, recurrent, or metastatic) according to international TNM staging; patients with highly suspected gene mutations or requiring reconfirmation of molecular pathological diagnosis; or patients previously treated at this institution who have obtained pathological samples and completed PDTF construction but have progressed to refractory tumors.
3. At least one measurable lesion according to RECIST v1.1 criteria; the lesion is expected to be sufficiently large (diameter greater than 2 cm), such that tissue collection does not affect pathological diagnosis or other clinical treatment needs, and residual tissue samples from pathological testing can be used to construct the PDTF model.
4. No prior systemic treatment, or disease progression or recurrence more than 6 months after previous neoadjuvant/adjuvant chemotherapy.
5. ECOG performance status of 0-1, ensuring the patient can tolerate biopsy and treatment.
6. Expected survival of at least 3 months, with no severe concomitant diseases affecting trial participation.
7. Adequate organ function, including:

   * Bone marrow function: Hemoglobin ≥80 g/L; Neutrophil count ≥1.5×10^9/L; White blood cell count ≥3.5×10^9/L; Platelet count ≥100×10^9/L;
   * Liver function: Serum total bilirubin ≤1.5×upper limit of normal (ULN); Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤3×ULN, or ≤5×ULN in patients with liver metastases;
   * Renal function: Serum creatinine ≤1.5×ULN, or creatinine clearance (CrCl) ≥60 mL/min (calculated using the Cockcroft-Gault formula);
   * Cardiac function: New York Heart Association (NYHA) classification < III; Left ventricular ejection fraction (LVEF) ≥50%.
8. Women of childbearing potential must use reliable contraception or have a negative pregnancy test (serum or urine) within 7 days prior to enrollment, and be willing to use appropriate contraception during the trial and for 8 weeks after the last dose of the study drug. Men must also agree to use appropriate contraception during the trial and for 8 weeks after the last dose of the study drug.
9. Voluntary participation in the study, signed informed consent form, good compliance, and willingness to cooperate with follow-up, including providing biological samples for PDTF construction and future research.

Exclusion Criteria

Patients meeting any of the following criteria are ineligible for enrollment. Exclusion criteria must be fully assessed during the screening period to ensure patient safety and the reliability of trial data.

1. No lesions available for biopsy, or concurrent or metachronous multiple primary malignant tumors, to avoid interference with efficacy evaluation.
2. Severe dysfunction of liver, kidney, heart, or other vital organs (e.g., Child-Pugh class C liver failure, NYHA class III-IV heart failure, creatinine clearance <30 mL/min).
3. Poor compliance, or contraindications to chemotherapy, targeted drugs, or immunotherapy (e.g., history of severe allergies); allergy to any study drug or its excipients, severe allergy history, or contraindications to the study drug.
4. Uncontrolled cardiovascular or cerebrovascular events, such as: NYHA class ≥2 heart failure; unstable angina; myocardial infarction within 1 year; clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; cerebral hemorrhage or infarction (excluding asymptomatic lacunar infarcts not requiring treatment); severe cardiovascular or cerebrovascular events within 12 months; uncontrolled hypertension (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg despite monotherapy); history of arterial thrombosis or deep vein thrombosis within 6 months prior to enrollment, or history of bleeding tendency or bleeding within 2 months prior to enrollment, regardless of severity; stroke or transient ischemic attack within 12 months prior to enrollment.
5. Active infection, uncontrolled hypertension, psychiatric disorders, or any condition that may affect trial safety/efficacy; severe chronic or active infections requiring systemic antibacterial, antifungal, or antiviral treatment, including tuberculosis (patients with a history of active tuberculosis ≥1 year prior to screening should also be excluded unless there is evidence of completed appropriate treatment); interstitial lung disease, noninfectious pneumonia, pulmonary fibrosis, history of acute lung disease, or poorly controlled systemic diseases (including but not limited to diabetes, hypertension); history of active immunodeficiency or autoimmune disease, including positive HIV test, other acquired or congenital immunodeficiency diseases, organ transplantation, or autoimmune diseases.
6. Presence of active brain metastases or leptomeningeal metastases.
7. Clinically significant pleural effusion, pericardial effusion, or ascites requiring drainage within 2 weeks prior to the first dose of the study drug.
8. Detectable second primary malignant tumor at enrollment, or history of other malignancies within the past 5 years (excluding adequately treated basal cell skin cancer or cervical carcinoma in situ).
9. Any major surgery within 28 days prior to the first dose of the study drug; history of allogeneic stem cell or organ transplantation.
10. Current gastrointestinal diseases, such as duodenal ulcer, ulcerative colitis, intestinal obstruction, or other conditions judged by the investigator as potentially leading to gastrointestinal bleeding or perforation; or history of unhealed intestinal perforation or fistula after surgical treatment.
11. Live vaccine received within 4 weeks prior to the first dose of the study drug (seasonal influenza vaccines are usually inactivated and thus allowed; intranasal vaccines are live and thus not allowed); receipt of herbal medicines or immunomodulatory drugs with anticancer indications (including thymosin, interferon, interleukin, except for local use to control ascites) within 2 weeks prior to the first dose of the study drug.
12. Pregnant or lactating women, or women of childbearing age not using effective contraception.
13. Current participation in other clinical trials, or recent (<4 weeks) experimental treatment; currently participating in interventional clinical research treatment, or receipt of other investigational drugs or use of investigational devices within 4 weeks prior to the first dose of the study drug.
14. Other factors judged by the investigator as potentially leading to early termination of the study, such as other serious diseases requiring concomitant treatment (including psychological or psychiatric disorders), significant laboratory abnormalities, or family or social factors that may affect patient safety or data and sample collection; other situations deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Until 3 months after the last patient is enrolled
  Proportion of patients achieving a best overall response of complete response (CR) or partial response (PR) according to RECIST v1.1 criteria. CR is defined as disappearance of all target lesions and normalization of tumor markers. PR is defined as at least a 30% decrease in the sum of diameters of target lesions compared with baseline.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Until 3 months after the last patient is enrolled
  Proportion of patients whose best overall response is complete response (CR), partial response (PR), or stable disease (SD) according to RECIST v1.1. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD).
Progression-Free Survival (PFS) | Until 12 months after the last patient is enrolled
  Time from first dose of PDTF-guided treatment to the first documented disease progression per RECIST v1.1 or death from any cause, whichever occurs first.
Feasibility of PDTF-Guided Treatment | Until 1 month after the last patient is enrolled
  Percentage of patients for whom PDTF model establishment and drug screening are successfully completed
Time to PDTF-Guided Treatment | Until 1 month after the last patient is enrolled
  Time from receipt of tumor tissue to finalization of a PDTF-guided treatment recommendation
Treatment-Related Adverse Events | Until 12 months after the last patient is enrolled
  Number and percentage of patients experiencing treatment-related adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE, 5.0). Adverse events will be summarized by type, frequency, and severity (Grade 1-5).
Biopsy-Related Complications | Until 12 months after the last patient is enrolled
  Number and percentage of patients experiencing complications related to tumor biopsy procedures performed for PDTF model establishment (e.g., bleeding, infection, pain requiring intervention, pneumothorax, or other procedure-related adverse events), graded using NCI CTCAE 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong Univertisy, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No